CLINICAL TRIAL: NCT01533922
Title: A Randomised, Double-blind, 5 Treatment Arms, 4-period, Incomplete Cross-over Study to Determine the Effect of 6 Weeks Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (FDC) (2.5 / 5 µg; and 5 / 5 µg) (Delivered by the Respimat® Inhaler) Compared With Tiotropium (5 µg), Olodaterol (5 µg ) and Placebo (Delivered by the Respimat® Inhaler) on Lung Hyperinflation and Exercise Endurance Time During Constant Work Rate Cycle Ergometry in Patients With Chronic Obstructive Pulmonary Disease (COPD) [MORACTO TM 1]
Brief Title: Effect on Exercise Endurance and Lung Hyperinflation of Tiotropium + Olodaterol in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.13; 2011-004659-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol; tiotropium-olodaterol

ARMS (5):
- Tiotropium + olodaterol High dose QD (Experimental): patient will receive tiotropium 5 mcg + olodaterol 5 mcg in a fixed dose combination once daily
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- Tiotropium + olodaterol Low dose QD (Experimental): patient will receive tiotropium 2.5 mcg + olodaterol 5 mcg in a fixed dose combination once daily
  Interventions: Drug: Tiotropium + Olodaterol; Device: Respimat
- Tiotropium 5 mcg QD (Active Comparator): patient will receive tiotropium 5 mcg once daily
  Interventions: Drug: Tiotropium; Device: Respimat
- Olodaterol 5 mcg QD (Active Comparator): patient will receive olodaterol 5 mcg once daily
  Interventions: Drug: Olodaterol; Device: Respimat
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Respimat

INTERVENTIONS:
Drug: Placebo — placebo matching tiotropium + olodaterol FDC
  Arms: Placebo QD
Drug: Tiotropium — Tiotropium 5 mcg once daily
  Arms: Tiotropium 5 mcg QD
Drug: Olodaterol — Olodaterol 5 mcg once daily
  Arms: Olodaterol 5 mcg QD
Drug: tiotropium + olodaterol — tiotropium + olodaterol 5 mcg once daily
  Arms: Tiotropium + olodaterol High dose QD
Drug: Tiotropium + Olodaterol — Tiotropium 2.5 mcg + Olodaterol 5 mcg once daily
  Arms: Tiotropium + olodaterol Low dose QD
Device: Respimat — Respimat inhaler

SUMMARY:
The primary objective of this trial is to investigate the effect of 6 weeks treatment with tiotropium + olodaterol fixed dose combination inhalation solution on lung hyperinflation and exercise tolerance in patients with COPD

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with a post-bronchodilator FEV1 <80% of predicted normal and a post-bronchodilator FEV1/FVC <70% at Visit 1.
3. Male or female patients, between 40 and 75 years of age (inclusive) on day of signing informed consent.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years.

Exclusion criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT >x2 ULN, SGPT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN will be excluded regardless of clinical condition
3. Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma.

   Patients with any of the following conditions:
4. A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists)
5. A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists)
6. A history of myocardial infarction within 1 year of screening visit (Visit 1)
7. Unstable or life-threatening cardiac arrhythmia
8. Hospitalized for heart failure within the past year
9. Known active tuberculosis
10. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed)
11. A history of life-threatening pulmonary obstruction
12. A history of cystic fibrosis
13. Clinically evident bronchiectasis
14. A history of significant alcohol or drug abuse
15. Any contraindications for exercise testing.
16. Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1)
17. Patients being treated with any oral ß-adrenergics
18. Patients being treated with oral corticosteroid medication at unstable doses
19. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
20. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program
21. Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnoea, such as arthritis in the leg, angina pectoris or claudication or morbid obesity.
22. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit
23. Patients with known hypersensitivity to ß-adrenergics drugs, anticholinergic drugs, BAC, EDTA or any other component of the Respimat® inhalation solution delivery system
24. Pregnant or nursing women
25. Women of childbearing potential not using highly effective methods of birth control.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (44):
- United States (8):
  - 1237.13.01302 Boehringer Ingelheim Investigational Site, Torrance, California
  - 1237.13.01308 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1237.13.01304 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1237.13.01307 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1237.13.01305 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1237.13.01301 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.13.01303 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.13.01306 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Argentina (2):
  - 1237.13.54301 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1237.13.54302 Boehringer Ingelheim Investigational Site, Mar del Plata
- Australia (5):
  - 1237.13.61306 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1237.13.61301 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1237.13.61305 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1237.13.61304 Boehringer Ingelheim Investigational Site, Footscray, Victoria
  - 1237.13.61302 Boehringer Ingelheim Investigational Site, Prahran, Victoria
- Austria (2):
  - 1237.13.43303 Boehringer Ingelheim Investigational Site, Linz
  - 1237.13.43301 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
- Belgium (5):
  - 1237.13.32302 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.13.32303 Boehringer Ingelheim Investigational Site, Edegem
  - 1237.13.32305 Boehringer Ingelheim Investigational Site, Jambes
  - 1237.13.32304 Boehringer Ingelheim Investigational Site, Lanaken
  - 1237.13.32301 Boehringer Ingelheim Investigational Site, Leuven
- Canada (3):
  - 1237.13.11302 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1237.13.11303 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 1237.13.11304 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Chile (2):
  - 1237.13.56301 Boehringer Ingelheim Investigational Site, Chile
  - 1237.13.56302 Boehringer Ingelheim Investigational Site, Santiago
- Germany (6):
  - 1237.13.49302 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.13.49307 Boehringer Ingelheim Investigational Site, Dortmund
  - 1237.13.49304 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.13.49301 Boehringer Ingelheim Investigational Site, Halle
  - 1237.13.49303 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.13.49305 Boehringer Ingelheim Investigational Site, Lübeck
- Italy (9):
  - 1237.13.39302 Boehringer Ingelheim Investigational Site, Genova
  - 1237.13.39304 Boehringer Ingelheim Investigational Site, Parma
  - 1237.13.39303 Boehringer Ingelheim Investigational Site, Pavia
  - 1237.13.39305 Boehringer Ingelheim Investigational Site, Pavullo Nel Frignano (mo)
  - 1237.13.39301 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.13.39312 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.13.39310 Boehringer Ingelheim Investigational Site, Roma
  - 1237.13.39308 Boehringer Ingelheim Investigational Site, Sesto S. Giovanni (mi)
  - 1237.13.39306 Boehringer Ingelheim Investigational Site, Trieste
- New Zealand (2):
  - 1237.13.64302 Boehringer Ingelheim Investigational Site, Christchurch
  - 1237.13.64301 Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ

REFERENCES:
- [Derived] O'Donnell DE, Casaburi R, Frith P, Kirsten A, De Sousa D, Hamilton A, Xue W, Maltais F. Effects of combined tiotropium/olodaterol on inspiratory capacity and exercise endurance in COPD. Eur Respir J. 2017 Apr 19;49(4):1601348. doi: 10.1183/13993003.01348-2016. Print 2017 Apr. PMID 28424359

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, 4-period incomplete block cross-over trial. 295 patients were randomized to one of five treatments sequences and treated. It was a double-blind trial in which each treatment period lasted 6 weeks with a washout period of 21 days between each.
Groups:
- Tio+Olo 2.5/5 / Tio+Olo 5/5 / Tio / Olo: Patients received a total of four treatments, and each treatment period is separated by a washout period of 21 days. The treatments administered orally via the respimat inhaler, once daily, in the morning were:
  * Fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
  * Tiotropium fixed dose 5 µg
  * Olodaterol fixed dose 5 µg
- Tio+Olo 5/5 / Tio / Olo / Placebo: Patients received a total of four treatments, and each treatment period is separated by a washout period of 21 days. The treatments administered orally via the respimat inhaler, once daily, in the morning were:
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
  * Tiotropium fixed dose 5 µg
  * Olodaterol fixed dose 5 µg
  * Oral inhalation of placebo
- Tio / Olo / Placebo / Tio+Olo 2.5/5: Patients received a total of four treatments, and each treatment period is separated by a washout period of 21 days. The treatments administered orally via the respimat inhaler, once daily, in the morning were:
  * Tiotropium fixed dose 5 µg
  * Olodaterol fixed dose 5 µg
  * Oral inhalation of placebo
  * Fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg
- Olo / Placebo / Tio+Olo 2.5/5 / Tio+Olo 5/5: Patients received a total of four treatments, and each treatment period is separated by a washout period of 21 days. The treatments administered orally via the respimat inhaler, once daily, in the morning were:
  * Olodaterol fixed dose 5 µg
  * Oral inhalation of placebo
  * Fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
- Placebo / Tio+Olo 2.5/5 / Tio+Olo 5/5 / Tio: Patients received a total of four treatments, and each treatment period is separated by a washout period of 21 days. The treatments administered orally via the respimat inhaler, once daily, in the morning were:
  * Oral inhalation of placebo
  * Fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
  * Tiotropium fixed dose 5 µg
Period: Overall Study
Arm/Group | Tio+Olo 2.5/5 / Tio+Olo 5/5 / Tio / Olo | Tio+Olo 5/5 / Tio / Olo / Placebo | Tio / Olo / Placebo / Tio+Olo 2.5/5 | Olo / Placebo / Tio+Olo 2.5/5 / Tio+Olo 5/5 | Placebo / Tio+Olo 2.5/5 / Tio+Olo 5/5 / Tio
Started | 59 | 59 | 60 | 58 | 59
Received Placebo | 0 | 49 | 57 | 57 | 59
Received Olo 5 | 51 | 52 | 57 | 57 | 0
Received Tio 5 | 54 | 58 | 59 | 1 (One patient received Tio 5 instead of Olo 5 by mistake.) | 54
Received Tio+Olo 2.5/5 | 59 | 0 | 52 | 55 | 56
Received Tio+Olo 5/5 | 58 | 59 | 0 | 53 | 56
Completed | 49 (Completed all treatment arms) | 47 (Completed all treatment arms) | 50 (Completed all treatment arms) | 53 (Completed all treatment arms) | 53 (Completed all treatment arms)
Not Completed | 10 | 12 | 10 | 5 | 6
Not completed — Adverse Event | 5 | 8 | 6 | 3 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 2 | 1
Not completed — Other reason not defined above | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) : This patient set included all patients of the Randomised Set (RS : patients who signed the informed consent form and were also randomised, regardless of whether the patient was treated with study medication or not) who were dispensed study medication and were documented to have taken at least 1 dose of study medication.
Groups:
- Overall Study: A randomised, double-blind, placebo controlled, 5 treatment, 4-period, incomplete, crossover study. Each treatment period was separated by a washout period of 21 days. The 5 treatments, administered orally via the respimat inhaler, once daily, in the morning were:
  * Oral inhalation of placebo
  * Olodaterol fixed dose 5 µg
  * Tiotropium fixed dose 5 µg
  * Fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg
  Treatment sequence is not considered as a factor which may affect the treatment effect due to sufficient washout period added between treatment cycles. As a result, we only display baseline characteristics as a whole population, but not by treatment sequence
Arm/Group | Overall Study
Number analyzed (Participants) | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 213

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Capacity at Rest Before Constant Work Rate Cycle Ergometry to Symptom Limitation at 75% Wcap
Description: Inspiratory capacity (IC) at rest before constant work rate cycle ergometry to symptom limitation at 75% maximal work capacity (Wcap).
  Wcap was defined as the maximum work rate achieved for at least 30 seconds during the incremental cycle ergometry performed at Visit 1.
  The presented means are adjusted means from the MMRM (Mixed Effects Model Repeated Measures) model.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS) : This patient set included all patients in the TS who had the study baseline and at least 1 evaluable post-dose measurement for 1 of the primary endpoints. Assignment to the FAS was done after implementation of any data handling rules,which set measurements to missing.
Measure: Mean (Standard Error); unit: Litres
Groups:
- Placebo: Oral inhalation of placebo, 2 puffs from the Respimat inhaler, once daily, in the morning.
- Olodaterol 5 µg: Oral inhalation of Olodaterol fixed dose 5 µg (2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium 5 µg: Oral inhalation of Tiotropium fixed dose 5 µg (2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium + Olodaterol 2.5/5: Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 µg and Olodaterol 5 µg (Tiotropium: 1.25 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium + Olodaterol 5/5: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
Arm/Group | Placebo | Olodaterol 5 µg | Tiotropium 5 µg | Tiotropium + Olodaterol 2.5/5 | Tiotropium + Olodaterol 5/5
Number analyzed (Participants) | 211 | 214 | 213 | 214 | 219
Litres | 2.440 (0.027) | 2.566 (0.027) | 2.571 (0.027) | 2.658 (0.027) | 2.685 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.244, 95% CI 2-sided [0.191 to 0.298], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 5/5 once daily (QD) minus Placebo
Statistical Analysis 2: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.119, 95% CI 2-sided [0.065 to 0.172], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Olodaterol 5 mcg
Statistical Analysis 3: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.061 to 0.167], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Tiotropium 5 mcg QD
Statistical Analysis 4: Comparison: Placebo vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.218, 95% CI 2-sided [0.164 to 0.271], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Placebo QD
Statistical Analysis 5: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 0.092, 95% CI 2-sided [0.038 to 0.145], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Olodaterol 5 mcg QD
Statistical Analysis 6: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.034 to 0.141], Standard Error of Mean 0.027 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Tiotropium 5 mcg QD

2. Primary Outcome: Endurance Time During Constant Work Rate Cycle Ergometry to Symptom Limitation at 75% Wcap
Description: Endurance time during constant work rate cycle ergometry (CWRCE) to symptom limitation at 75% work capacity (Wcap).
  Wcap was defined as the maximum work rate achieved for at least 30 seconds during the incremental cycle ergometry performed at Visit 1.
  The presented means are adjusted mean from the MMRM model.
Time Frame: 6 weeks
Population: FAS
Measure: Geometric Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Olodaterol 5 µg | Tiotropium 5 µg | Tiotropium + Olodaterol 2.5/5 | Tiotropium + Olodaterol 5/5
Number analyzed (Participants) | 209 | 208 | 209 | 212 | 212
seconds | 375.45 (12.037) | 453.38 (14.552) | 457.16 (14.652) | 474.80 (15.145) | 454.08 (14.474)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Ratio = 1.209, 95% CI 2-sided [1.132 to 1.292], Standard Error of Mean 0.041 — Ratio calculated as Tiotropium + olodaterol 5/5 QD divided by Placebo QD
Statistical Analysis 2: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p = 0.9633, Mixed Models Analysis; Ratio = 1.002, 95% CI 2-sided [0.937 to 1.070], Standard Error of Mean 0.034 — Ratio calculated as Tiotropium + olodaterol 5/5 QD divided by Olodaterol 5 mcg QD
Statistical Analysis 3: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p = 0.8415, Mixed Models Analysis; Ratio = 0.993, 95% CI 2-sided [0.930 to 1.061], Standard Error of Mean 0.033 — Ratio calculated as Tiotropium + olodaterol 5/5 QD divided by Tiotropium 5 mcg QD
Statistical Analysis 4: Comparison: Placebo vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Ratio = 1.265, 95% CI 2-sided [1.184 to 1.351], Standard Error of Mean 0.042 — Ratio calculated as Tiotropium + olodaterol 2.5/5 QD divided by Placebo QD
Statistical Analysis 5: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.1717, Mixed Models Analysis; Ratio = 1.047, 95% CI 2-sided [0.980 to 1.119], Standard Error of Mean 0.035 — Ratio calculated as Tiotropium + olodaterol 2.5/5 QD divided by Olodaterol 5 mcg QD
Statistical Analysis 6: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.2610, Mixed Models Analysis; Ratio = 1.039, 95% CI 2-sided [0.972 to 1.110], Standard Error of Mean 0.035 — Ratio calculated asTiotropium + olodaterol 2.5/5 QD divided by Tiotropium 5 mcg QD

3. Secondary Outcome: Slope of the Intensity of Breathing Discomfort During Constant Work Rate Cycle Ergometry to Symptom Limitation at 75% Work Capacity
Description: Slope of the intensity of breathing discomfort during Constant Work Rate Cycle Ergometry (CWRCE) to symptom limitation at 75% Work capacity (Wcap). The intensity of breathing discomfort was rated using the modified Borg scale with ratings from 0 (nothing at all) to 10 (maximal).
  Slope of breathing discomfort is defined as: (intensity of breathing discomfort at the end of exercise minus intensity of breathing discomfort at rest) / endurance time.
  A decrease in slope indicates improvement.
  The presented means are adjusted means from MMRM model.
Time Frame: 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale / second
Arm/Group | Placebo | Olodaterol 5 µg | Tiotropium 5 µg | Tiotropium + Olodaterol 2.5/5 | Tiotropium + Olodaterol 5/5
Number analyzed (Participants) | 209 | 208 | 209 | 212 | 212
units on a scale / second | 0.018 (0.001) | 0.016 (0.001) | 0.016 (0.001) | 0.015 (0.001) | 0.016 (0.001)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.004 to -0.001], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Placebo QD
Statistical Analysis 2: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p = 0.8291, Mixed Models Analysis; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [-0.001 to 0.002], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Olodaterol 5 mcg QD
Statistical Analysis 3: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p = 0.8570, Mixed Models Analysis; Mean Difference (Final Values) = -0.000, 95% CI 2-sided [-0.002 to 0.001], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Tiotropium 5 mcg QD
Statistical Analysis 4: Comparison: Placebo vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.005 to -0.002], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Placebo QD
Statistical Analysis 5: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.7294, Mixed Models Analysis; Mean Difference (Final Values) = -0.000, 95% CI 2-sided [-0.002 to 0.001], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Olodaterol 5 mcg QD
Statistical Analysis 6: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p = 0.4567, Mixed Models Analysis; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.002 to 0.001], Standard Error of Mean 0.001 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Tiotropium 5 mcg QD

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (One Hour Post-dose)
Description: Forced Expiratory Volume in 1 Second (FEV1) (one hour post-dose)
  The presented means are adjusted means from MMRM model.
Time Frame: 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo | Olodaterol 5 µg | Tiotropium 5 µg | Tiotropium + Olodaterol 2.5/5 | Tiotropium + Olodaterol 5/5
Number analyzed (Participants) | 216 | 214 | 218 | 216 | 224
Litres | 1.497 (0.013) | 1.689 (0.013) | 1.706 (0.013) | 1.783 (0.013) | 1.820 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.323, 95% CI 2-sided [0.293 to 0.352], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Placebo QD
Statistical Analysis 2: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [0.101 to 0.160], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Olodaterol 5 mcg QD
Statistical Analysis 3: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.084 to 0.143], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 5/5 QD minus Tiotropium 5 mcg QD
Statistical Analysis 4: Comparison: Placebo vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.286, 95% CI 2-sided [0.256 to 0.315], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Placebo QD
Statistical Analysis 5: Comparison: Olodaterol 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [0.063 to 0.123], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Olodaterol 5 mcg QD
Statistical Analysis 6: Comparison: Tiotropium 5 µg vs Tiotropium + Olodaterol 2.5/5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.047 to 0.106], Standard Error of Mean 0.015 — Difference calculated as Tiotropium + olodaterol 2.5/5 QD minus Tiotropium 5 mcg QD

ADVERSE EVENTS:
Time Frame: From drug administration until 21 days after the last administration, up to 120 days
Arm/Group | Placebo | Olodaterol 5 µg | Tiotropium 5 µg | Tiotropium + Olodaterol 2.5/5 | Tiotropium + Olodaterol 5/5
Serious Adverse Events (participants affected / at risk) | 4/222 | 3/217 | 8/226 | 5/222 | 6/226
Other Adverse Events (participants affected / at risk) | 26/222 | 17/217 | 20/226 | 13/222 | 19/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Olodaterol 5 µg (N=217) | Tiotropium 5 µg (N=226) | Tiotropium + Olodaterol 2.5/5 (N=222) | Tiotropium + Olodaterol 5/5 (N=226)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Olodaterol 5 µg (N=217) | Tiotropium 5 µg (N=226) | Tiotropium + Olodaterol 2.5/5 (N=222) | Tiotropium + Olodaterol 5/5 (N=226)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 26 | 17 | 20 | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.